CLINICAL TRIAL: NCT06905730
Title: Minimal Clinically Important Difference (MCID) of Clinical Test of Sensory Interaction on Balance (CTSIB) in Individuals With Sub-Acute Stroke
Brief Title: Minimal Clinically Important Difference of Clinical Test of Sensory Interaction on Balance in Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/790
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sensory integration deficits in balance
  Interventions: Diagnostic Test: sensory integration deficits in balance

INTERVENTIONS:
Diagnostic Test: sensory integration deficits in balance — By assessing sensory integration deficits in balance recovery, the study will help establish meaningful thresholds for rehabilitation outcomes, guiding clinicians in tailoring therapy for improved post-stroke balance and functional independence

SUMMARY:
"Stroke is a major cause of disability worldwide, often leading to balance impairments due to deficits in sensory integration and motor control. These impairments hinder postural stability and functional independence, making balance rehabilitation a critical focus in sub-acute stroke care.

DETAILED DESCRIPTION:
The objective of this study is to determine the Minimal Clinically Important Difference (MCID) for the Clinical Test of Sensory Interaction on Balance (CTSIB) in individuals with sub-acute stroke rehabilitation. CTSIB evaluates the sensory contributions (visual, vestibular, and somatosensory) to balance by testing an individual's ability to maintain stability under various conditions. Additionally, the Berg Balance Scale (BBS) will be used to assess functional balance, and the Global Rating of Change (GRC) will be included as a subjective measure to gauge participants' perceived improvement in balance and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Type of stroke Participants must have experienced a first unilateral hemispheric supratentorial stroke, which may be either ischemic or hemorrhagic in nature.
* Only individuals who have been clinically diagnosed with a stroke within the past 3 to 6 months will be included.
* Participants must have a Functional Ambulation Classification (FAC) score of 3, indicating independent ambulation with supervision or the use of a walking aid.
* The individual must have sufficient cognitive and communication abilities to understand and follow instructions during assessments.
* The study will include patients in the early subacute phase of stroke recovery, defined as 7 days to 3 months post-onset.
* Participants must have a Montreal Cognitive Assessment (MoCA) score of at least 24, indicating normal cognitive function or only mild cognitive impairment

Exclusion Criteria:

* Individuals with severe cognitive impairments that prevent them from understanding, consenting to, or following simple instructions will be excluded.
* Participants with uncontrolled medical conditions such as cardiovascular disease or uncontrolled diabetes will not be eligible for the study.
* Individuals diagnosed with nerve compression conditions affecting motor or sensory function will be excluded.
* Patients exhibiting significant hemispatial neglect following a stroke will not be included in the study.
* Participants showing signs of unilateral spatial neglect, impacting their ability to process stimuli on one side, will be excluded.
* Patients who test positive for unilateral spatial neglect using the Catherine Line Bisection Test will be excluded.
* Individuals with severe visual impairments that compromise independent ambulation will not be eligible.
* Patients with gait disturbances due to conditions other than stroke (e.g., Parkinson's disease, severe arthritis) will be excluded.
* Individuals who are unable to comply with study protocols or behavioral requirements will not be included.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Difference of Clinical Test of Sensory Interaction on Balance in Individuals Withhaving a Montreal Cognitive Assessment (MoCA) score of at least 24, indicating normal cognitive function or only mild cognitive impairment.
  Participants must have a Functional Ambulation Classification (FAC) score of 3, indicating independent ambulation with supervision or the use of a walking aid.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 12 Months
  Berg balance scale scores range from 0 to 56. The lower your score, the more at risk you are for losing your balance. The higher your score, the better your functional mobility (ability to move effectively and safely)
Functional Ambulation Classification (FAC): | 12 Months
  The Functional Ambulation Classification (FAC) is a tool used to assess and categorize functional mobility and gait in patients, ranging from non-functional ambulation (0) to independent ambulation (5), quantifying levels of assistance, supervision, and limited mobility.
Global Rating of Change (GRC) | 12 Months
  The Global Rating of Change (GRC) scale is a tool used to assess a patient's perceived improvement or deterioration over time, typically following treatment, on a scale ranging from "a very great deal worse" (-7) to "a very great deal better" (+7), with 0 indicating "no change

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No